CLINICAL TRIAL: NCT06698289
Title: Prevalence of Preoperative Sarcopenia and Its Impact on Surgical Outcomes in Patients With Colorectal Cancer: A Prospective Study
Brief Title: Preoperative Sarcopenia and Surgical Outcomes in Colorectal Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hilmi Bozkurt, Associate Professor, Mersin University
Other Study IDs: CRC-SARCOPENIA-MUNIV2024
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Colon Cancer; Rectal Cancer; Surgical Outcomes
MeSH Terms: conditions — Sarcopenia; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia: Patients who meet the diagnostic criteria for sarcopenia will be included in this group. The diagnosis of sarcopenia will be made using the criteria defined by the European Working Group on Sarcopenia in Older People (EWGSOP). This requires the presence of both low muscle strength (e.g. low handgrip strength) and low muscle quantity/quality (e.g. low skeletal muscle index on CT scan). Patients will further classified into stages of "probable sarcopenia", "sarcopenia", and "severe sarcopenia" based on the severity.
- Non-sarcopenia: Patients who do not meet the diagnostic criteria for sarcopenia will be included in this group. They will have normal or above-normal muscle strength and muscle quantity/quality measurements. This group will serve as the comparison cohort to evaluate the impact of sarcopenia on surgical outcomes.

SUMMARY:
Colorectal cancer is the third most common malignant neoplasm worldwide and the fourth leading cause of cancer-related deaths. Muscle mass loss in oncology patients is most often the result of cancer-related malnutrition.

Sarcopenia is a progressive and generalized skeletal muscle disorder associated with increased likelihood of adverse outcomes such as physical disability, poor quality of life, and death. It is characterized by low muscle strength, low muscle quantity and quality, and low physical performance. Sarcopenia is highly prevalent in older adults and those with chronic diseases, including cancer. In the context of colorectal cancer, preoperative sarcopenia has been linked to increased postoperative complications, longer hospital stays, and reduced survival.

The aim of this prospective observational study is to evaluate the prevalence of preoperative sarcopenia and postoperative outcomes in patients with colorectal cancer, using validated methods to assess muscle strength, muscle mass, and physical performance.

DETAILED DESCRIPTION:
Sarcopenia is directly responsible for functional impairment in the body, increased risk of falls, loss of autonomy, decreased respiratory capacity, and reduced immunity. The diagnostic criteria for sarcopenia include three main components: reduced muscle strength, low muscle quantity, and poor physical performance. Based on these criteria, sarcopenia is categorized into three stages: probable sarcopenia, sarcopenia, and severe sarcopenia.

The relationships between sarcopenia and poor prognosis, such as high postoperative mortality, chemotherapy toxicity, reduced survival, increased infection rates, and prolonged hospital stays, have been emphasized. Surgical resection is an important aspect of colorectal cancer management, and the assessment of sarcopenia as a predictor of perioperative or postoperative morbidity risk can provide valuable prognostic information for surgeons and patients. Therefore, patients diagnosed with colorectal cancer should be screened for sarcopenia from the beginning of their treatment, informed about the potential adverse effects of sarcopenia, and the importance of sarcopenia prevention and treatment strategies should be emphasized.

The prevalence and impact of sarcopenia in patients with colorectal cancer are not well known, as most studies have classified sarcopenia solely based on the presence of low muscle mass on CT scans, which may overestimate the prevalence. The aim of this prospective observational study is to evaluate the prevalence of preoperative sarcopenia and its impact on postoperative outcomes in patients with colorectal cancer, by combining 5 different test methods defined by the European Working Group on Sarcopenia in Older People (EWGSOP) to assess muscle strength, muscle mass, and physical performance. These test are:

* SARC-F Questionnaire: The SARC-F is a 6-item questionnaire used as a screening tool for sarcopenia. It evaluates 5 components: Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls. Each component is scored from 0 to 2, with a total score ranging from 0 to 10. A score of 4 or higher is considered indicative of sarcopenia.
* Handgrip Strength Test: Handgrip strength is a proxy measure for overall muscle strength. It is measured using a hand-held dynamometer, with the patient sitting or standing and the arm positioned at a 90-degree angle. Patients perform the test twice, and the higher of the two measurements is recorded. Handgrip strength thresholds for sarcopenia diagnosis: Men: <27 kg, Women: <16 kg
* 4-Meter Gait Speed Test: This test measures the time it takes a patient to walk 4 meters at their usual pace. Patients start from a standing position and walk at their normal comfortable speed. The time taken to complete the 4-meter distance is recorded. Gait speed threshold for sarcopenia diagnosis: <0.8 m/s
* 5-Times Sit-to-Stand Test: This test evaluates lower extremity muscle strength and function. Patients start from a seated position in a standard chair, then fully stand up and sit back down 5 times as quickly as possible. The time taken to complete the 5 repetitions is recorded. Threshold for sarcopenia diagnosis: 15 seconds
* Muscle Measurement on Preoperative CT Scans: CT scans performed for diagnostic or staging purposes are used to assess muscle mass. The cross-sectional area of skeletal muscle is measured at the third lumbar vertebra (L3) level. This L3 skeletal muscle area is normalized to the patient's height squared to calculate the Skeletal Muscle Index (SMI). Thresholds for sarcopenia based on SMI: Men: <43 cm²/m² , Women: <41 cm²/m²

By assessing these different parameters - self-reported function, muscle strength, gait speed, and muscle mass - the study can comprehensively evaluate the presence and severity of sarcopenia in the colorectal cancer patients. The combination of these validated tools provides a robust diagnosis of sarcopenia according to the EWGSOP criteria.

A power analysis was performed using the G*Power (v3.1.7) program to determine the sample size. The power of the study is expressed as 1-β (where β is the probability of a type II error). Based on the study by Ying Zhang et al. titled "Sarcopenia and Its Influencing Factors in Patients With Colorectal Cancer", the difference in grip strength measurements between the sarcopenia and non-sarcopenia groups was used for the calculation. The resulting effect size was calculated as d=0.901, and it was determined that a total of 64 participants, with at least 34 in each group, would be required to achieve 95% power at an α level of 0.05.

This study will include at least 64 patients who meet the inclusion and exclusion criteria. Patients with colorectal cancer who are admitted to the General Surgery Department of Mersin University Hospital and have an indication for surgical intervention will undergo the appropriate surgical procedure. The method to be applied is decided by discussing with the patient, based on the patient and the size of the disease.

The data for this study will be collected between November 2024, and November 2025. During this period, the data of patients who were operated on for colorectal cancer at the General Surgery Department in Mersin University Hospital will be collected. The patients' demographic characteristics, history of semptoms, height, weight, hand grip strength test, 4-meter walking test, 5-time sit-to-stand test, and preoperative computed tomography findings will be recorded at the first admission.

After the surgery, the surgical findings, examination findings, wound complications, and the time to return to daily life will be examined. This data will be obtained through the retrospective review of medical records and confirmed by face-to-face interviews with patients who have attended the outpatient clinic, and then recorded in the data collection form.

Data collection will continue until at least 32 patients each are reached in the sarcopenia and non-sarcopenia groups. Once the target sample size is reached, new data collection from patients will be terminated, and statistical analyses will be performed to compare the prevalence between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of colon cancer
* Having undergone surgery at Mersin University General Surgery Department as of 15.11.2024
* Patients aged 18 years and above
* Patients whose descriptive and clinical characteristics are recorded in their medical files
* Those who have signed the Informed Volunteer Consent Form/Written Consent Form

Exclusion Criteria:

* Patients under 18 years of age
* Patients whose descriptive and clinical characteristics are not recorded in the file records
* Those who did not sign the Informed Volunteer Form/Written Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will be conducted at the Department of General Surgery, Mersin University Hospital, between November 15, 2024, and November 15, 2025. The study population consists of adult patients (≥18 years) diagnosed with colorectal cancer who are scheduled for surgical intervention.
  Patients will be categorized into sarcopenia and non-sarcopenia groups based on EWGSOP criteria, incorporating muscle strength, muscle mass, and physical performance measurements.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 30 days post-surgery
  Postoperative complications will be systematically evaluated and graded according to the Clavien-Dindo Classification system over a 30-day follow-up period. All complications will be documented daily during hospitalization and at scheduled follow-up visits, with particular attention to surgical site infections, anastomotic leakage, pulmonary complications, and prolonged ileus. This comprehensive assessment will enable detailed analysis of the relationship between preoperative sarcopenia and postoperative outcomes, potentially identifying high-risk patients who might benefit from preoperative optimization strategies.

SECONDARY OUTCOMES:
Length of Hospital Stay | 30 days post-surgery
  The duration of hospitalization will be measured from the day of surgery until discharge, with standardized discharge criteria including adequate pain control, successful oral intake and return of bowel function
Return to Daily Activities | 30 days post-surgery
  The evaluation of the patients' return to their initial functional status will be evaluated using standardized questionnaires, either in person during outpatient clinic visits or over the phone (in cases where they do not come for regular follow-ups). This involves monitoring the time required to resume basic activities of daily living (ADLs) and reach preoperative functional capacity.
Wound Healing Assessment | 30 days post-surgery
  Comprehensive wound healing evaluation will be conducted using standardized assessment tools and objective measurements throughout the 30-day postoperative period. Markers of wound healing will include inflammatory markers (C-reactive protein, white blood cell count), tissue oxygenation assessment, and time to suture/staple removal. The relationship between preoperative sarcopenia and wound healing complications will be analyzed, particularly focusing on the impact of reduced muscle mass and potential nutritional deficiencies on tissue repair and regeneration processes.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Yılmaz, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data underlying the study's primary and secondary outcomes. This includes demographic information (age, gender, BMI), clinical parameters (tumor staging, histology), sarcopenia assessment data (SARC-F scores, grip strength, walking tests, CT measurements), surgical details, and postoperative outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months and ending 36 months following article publication. Data access will be granted to researchers who provide a methodologically sound proposal and have received approval from an independent review committee. Proposals should be directed to the General Surgery Department of Mersin University Hospital.
Access Criteria: To gain access, researchers will need to sign a data access agreement and obtain relevant ethics approval if required. The study protocol, statistical analysis plan, informed consent form, and clinical study report will also be made available. Data will be shared through a secure online platform, with appropriate privacy and security safeguards in place.